CLINICAL TRIAL: NCT05835752
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple-Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RAY1225
Brief Title: The Safety, Tolerability and Pharmacokinetic Study of RAY1225
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RAY1225-22-01
Record Dates: First submitted 2023-04-11; First posted 2023-04-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obese; Healthy
Keywords: obesity; GLP-1; GIP
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- RAY1225(Part A) (Experimental): Escalating doses of RAY1225 administered subcutaneously (SC) once in healthy participants.
  Interventions: Drug: RAY1225
- Placebo (Part A) (Experimental): Placebo administered SC once in healthy participants.
  Interventions: Drug: Placebo
- RAY1225 (Part B) (Experimental): Escalating doses RAY1225 administered SC once weekly for four weeks in healthy participants.
  Interventions: Drug: RAY1225
- Placebo (Part B) (Experimental): Placebo administered SC once weekly for four weeks in healthy participants.
  Interventions: Drug: Placebo
- RAY1225(Part C) (Experimental): Three dose levels of RAY1225 administered SC once weekly for four weeks in participants with Obese.
  Interventions: Drug: RAY1225
- Placebo (Part C) (Experimental): Placebo administered SC once weekly for four weeks in participants with Obese.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAY1225 — Administered SC
  Arms: RAY1225(Part A)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A)
Drug: RAY1225 — Administered SC
  Arms: RAY1225 (Part B)
Drug: Placebo — Administered SC
  Arms: Placebo (Part B)
Drug: RAY1225 — Administered SC
  Arms: RAY1225(Part C)
Drug: Placebo — Administered SC
  Arms: Placebo (Part C)

SUMMARY:
This trial is conducted in China. The aim of the trial is to investigate safety, tolerability, pharmacokinetics and pharmacodynamics of RAY1225

ELIGIBILITY:
Inclusion Criteria:

1. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.
2. Participants must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.
3. Participants (including partners) must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.
4. Body weight is no less than 50 kg in males and no less than 45 kg in females. Body mass index (BMI) 18≤BMI<28 kg/m2（Part A&B only);BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
5. BMI≥28 kg/m2（Part C only）.BMI is determined by the following equation: BMI = weight/height2 (kg/m2).

Exclusion Criteria:

1. Participants with clinically significant disorders (including but not limited to, cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immune, neurological, psychiatric, cutaneous, hematological disorders, retinopathy, and neoplasms etc. )within 24 weeks prior to randomization.
2. Participants who are not suitable for subcutaneous injections (trauma, surgery, allergies or skin lesions, etc.).
3. Known history of definite mental illness, such as depression, suicidal ideation, schizophrenia, bipolar disorder.
4. Have a family or personal history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia (MEN) Syndrome type 2 or with thyroid nodules of unknown etiology found at screening and considered clinically significant by the investigator.
5. Participants who experienced a grade 3 hypoglycemic event within the 12 months prior to randomization, or experienced a hypoglycemic event (venous or terminal blood glucose <3 mmol/L ) ≥3 times or with hypoglycemia-related symptoms within 3 months prior to randomization.
6. Participants with clinically significant abnormalities on ECG, or QTcF >450ms, or with a family history of long QT syndrome or a family history of Brugada syndrome.
7. Participants who planning to use glucagon-like peptide-1 (GLP-1) receptor agonists and GLP1-related drugs or other enteroglucagon peptides(including but not limited to: exenatide, liraglutide, lisnatide, benalutide, dulaglutide, lorcetide, semaglutide, tirzepatide), during the 12 weeks prior to randomization or during the trial.
8. Participants who undergone major surgery, donated blood/bleeding profusely (> 400 mL) 12 weeks prior to randomization, donated blood/bleeding profusely (>200 mL) 4 weeks prior to randomization,or have a serious infection.
9. The average daily smoking are more than 5 cigarettes within 12 weeks prior to screening or unwilling to quit smoking during the study period.
10. Participants who may not complete the study for other reasons or should not be included in the study in the opinion of the investigator.
11. Known presence of a single genetic mutation, other diseases or medications causing obesity, including but not limited to hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, insulinoma, growth hormone deficiency, acromegaly, pseudohypoparathyroidism, hypogonadism, or weight gain caused by increased non-fat content (e.g., edema)[Part C only]

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
Number and severity of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events(SAE) | Baseline through Day 29 (Part A)
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported
Number and severity of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events(SAE) | Baseline through Day 71 (Part B&C)
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported

SECONDARY OUTCOMES:
To determine the single oral dose pharmacokinetic profiles of RAY1225(AUC0-∞) | Baseline through Day 29 (Part A)
To determine the multiple oral dose pharmacokinetic profiles of RAY1225(AUC0-∞) | Baseline through Day 71(Part B&C)
To determine the Pharmacodynamics of RAY1225(Change in Body Weight） | Baseline through Day 71(Part C)
To determine the Pharmacodynamics of RAY1225（Change in Waist circumference） | Baseline through Day 71(Part C)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital,South Medical Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No